CLINICAL TRIAL: NCT06811805
Title: Post-Marketing Clinical Follow Up Study to Further Assess the Safety & Efficacy of RenalGuard® Therapy in the Prevention of Cardiac Surgery Associated Acute Kidney Injury (CSA-AKI)
Brief Title: Post-Marketing Study to Assess the Safety & Efficacy of RenalGuard® Therapy for Prevention CSA-AKI
Acronym: KIDNEY-II
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CardioRenal Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RG-CSA-002
Record Dates: First submitted 2025-01-22; First posted 2025-02-06 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: AKI - Acute Kidney Injury; Cardiac Surgery Associated - Acute Kidney Injury
Keywords: RenalGuard; AKI; Acute Kidney Injury; Cardiac Surgery Associated AKI; CSA-AKI; AKI Prevention; Cardiac Surgery
MeSH Terms: conditions — Acute Kidney Injury | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Standard of care
  Interventions: Other: Standard of Care (SOC)
- RenalGuard Therapy (Experimental): RenalGuard Therapy
  Interventions: Device: RenalGuard Therapy

INTERVENTIONS:
Device: RenalGuard Therapy — RenalGuard Therapy
  Arms: RenalGuard Therapy
Other: Standard of Care (SOC) — Standard of care
  Arms: Control

SUMMARY:
The goal of this clinical trial is to assess the effect of RenalGuard Therapy in reducing the rates of Acute Kidney Injury (AKI) within 72 hours after cardiac surgery in patients at risk of developing Cardiac Surgery Associated AKI (CSA-AKI) compared to standard-of-care (SoC).

Participants will be randomized (1:1) to one of the two study groups. The Treatment study group will be managed with the RenalGuard System. The RenalGuard treatment will start after induction of anesthesiology and will run during surgery and for 6-7 hours in the Intensive Care Unit (ICU). The treatment will aim to achieve a urine rate above a predefined urine rate threshold. Patients in the control group will be managed based on the usual clinical practice in cardiac surgery centres as detailed in the recommendations for CSA-AKI prevention by accepted clinical guidelines.

For both study groups general anaesthesia, cardiopulmonary bypass (CPB) run and overall patient care will be based on SoC for cardiac surgery.

Patients will be followed up for up to 7 days post surgery or until discharge, which ever comes first.

Long-term follow up will be performed at 90 days post surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female and >18 years of age
2. Patient able to give written consent
3. Scheduled for the following non-emergent cardiac surgery procedure requiring CPB, isolated or in combination:

   * coronary artery bypass graft (CABG)
   * aortic valve replacement or repair alone, with or without aortic root repair
   * mitral, tricuspid, or pulmonic valve replacement or repair
   * simultaneous replacement of several cardiac valves
   * CABG with aortic, mitral, tricuspid, or pulmonic valve replacement or repair
   * Surgery on the aorta: aortic root and/ or ascending aorta
   * Atrial fibrillation (AF) ablation surgery if combined with other cardiac procedures.
   * Atrial septal defect (ASD) closure if combined with other cardiac procedures.
   * Excision of myxoma if combined with other cardiac procedures
4. Have at least one of the following risk factors for CSA-AKI:

   * CKD-EPI eGFR 20-59 mL/min/1.73 m²
   * Age ≥ 75 years
   * Undergoing combined surgery (e.g. CABG + Valve)
   * Logistic EuroScore of ≥5 or, Euroscore II of ≥4 or Society of Thoracic Surgeons (STS) Score ≥4
   * Left ventricular ejection fraction (LVEF) ≤ 35% by invasive or noninvasive diagnostic cardiac imaging performed within 90 days prior to surgery.
   * Insulin-requiring diabetes
   * Non-insulin-requiring diabetes with HbA1C ≥ 6.1% in the last 6 months
   * Preoperative anemia within 4 weeks of surgery

Exclusion Criteria:

1. Patient requiring emergency surgery
2. Surgery to be performed without CPB
3. Patient receiving furosemide at a dose>100 mg/day orally (or the equivalent dose of an alternative loop diuretic) in the last week
4. Patient who cannot be urethrally catheterize for any reason
5. Patients already dialysis dependent
6. Patients with CKD-EPI eGFR <20 mL/min/1.73 m²
7. Known or suspected AKI (KDIGO criteria) at the time of screening
8. Patients participating in another interventional drug or device study or have received an investigational drug or device treatment within the last 30 days
9. Pregnant patient, self-reported
10. Patients whose planned surgery to be performed under conditions of circulatory arrest or hypothermia with rectal temperature < 28°Celsius (82.4° Fahrenheit)
11. Patient with suspected or confirmed bacteraemia, endocarditis, or pyelonephritis at hospital admission
12. Patients with pneumonia, aspiration, or bilateral pulmonary infiltrates from an infectious aetiology reported on chest x-ray or CT scan in the last 7 days
13. Patients in cardiogenic shock or hemodynamic instability which require inotropes or vasopressors or other mechanical devices (Impella Heart Pump, IABP) within 24 hours prior to surgery
14. Patients on extracorporeal membrane oxygenation (ECMO) or durable ventricular assist device (VAD) at the time of screening, or planned use within 24h prior to surgery
15. Patients currently treated with chemotherapy or radiation therapy that may have an impact on kidney function.
16. Patient underwent prior solid organ transplantation
17. Patients underwent major surgery within the last 3 months
18. Any condition which, in the judgement of the investigator, might increase the risk to the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-02-23 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
CSA-AKI incidence between study groups | Within 72 hours
  CSA-AKI is defined as when any of the following three criteria are met:
  1. An increase in serum creatinine (SCr) by ≥0.3 mg/dl (≥26.5 umol/l) within 72 hours compared to the baseline value; OR
  2. An increase in SCr by ≥1.5 times from SCr value at baseline within 72 hours; OR
  3. Use of Renal Replacement Therapy (RRT) within 7 days of surgery or by hospital discharge (whichever is the earliest)

SECONDARY OUTCOMES:
A composite safety endpoint which includes: Significant severe clinically meaningful change in electrolytes (K+, Mg+2, Na+), New onset of postoperative atrial fibrillation, and Pulmonary edema | Within 72 hours
CSA-AKI Stage | Within 72 hours
  CSA-AKI severity by stage distribution between the study groups
CSA-AKI Incidence | Within 7 days
  AKI incidence within 7 days based on the KDIGO definition described in the primary endpoint section
CSA-AKI Duration | Within 7 days
  Duration of AKI within 7 days of surgery

OTHER OUTCOMES:
The incidence of Major Adverse Kidney Events (MAKE) | 90 days post-surgery
  MAKE-90 will be defined as:
  * Death within 90 days
  * Any dialysis within 90 days
  * A decrease of 25% in Estimate glomerular filtration rate (eGFR) from baseline eGFR level at 90 days
ICU and in-hospital length of stay | 7 days
Cumulative costs of ICU stay | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Raphael, MD, Principal Investigator — Thomas Jefferson University Hospitals
Locations (8):
- Jessa Medica Center, Hasselt, Belgium
- Germany (2):
  - TUM Klinikum Deutsches Herzzentrum, Munich
  - Uniklinikum Munster, Münster
- Israel (2):
  - Rambam Medical Center, Haifa
  - Rabin Medical Center - Belinson Campus, Petah Tikva
- Spain (2):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication

REFERENCES:
- [Background] Luckraz H, Giri R, Wrigley B, Nagarajan K, Senanayake E, Sharman E, Beare L, Nevill A. Balanced forced-diuresis as a renal protective approach in cardiac surgery: Secondary outcomes of electrolyte changes. J Card Surg. 2021 Nov;36(11):4125-4131. doi: 10.1111/jocs.15925. Epub 2021 Aug 19. PMID 34414606
- [Background] Luckraz H, Giri R, Wrigley B, Nagarajan K, Senanayake E, Sharman E, Beare L, Nevill A. Reduction in acute kidney injury post cardiac surgery using balanced forced diuresis: a randomized, controlled trial. Eur J Cardiothorac Surg. 2021 Apr 13;59(3):562-569. doi: 10.1093/ejcts/ezaa395. PMID 33236105